CLINICAL TRIAL: NCT05880628
Title: Evaluation of Faisability, Safety and Effectiveness and of Discogel in Patients With Aneurysmal and Simple Bone Cysts
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN552022/CHUSTE
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Bone Cysts
Keywords: Bone Cysts; Aneurysmal Bone Cysts; simple Bone Cysts; Discogel; Effectiveness; Safety
MeSH Terms: conditions — Bone Cysts; Bone Cysts, Aneurysmal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Any patient with aneurysmal or simple bone cyst who benefit a sclerotherapy by Discogel®: Any patient with aneurysmal or simple bone cyst who benefit a sclerotherapy by Discogel® will be included.
  Analysis datas of medical record.
  Interventions: Other: datas of medical record.

INTERVENTIONS:
Other: datas of medical record. — Analysis datas of medical record:
  * Feasibility of the technique
  * Safety of the technique
  * Efficacity (sclerose of the lesion)

SUMMARY:
There is no consensus in the scientific literature for the treatment of aneurysmal and simple bone cysts. Some scientific articles with utilisation of sclerosis agents for the treatment of aneurysmal bone cysts: Ethibloc no longer marketed, pure Ethanol, Aetoxisclerol.

DETAILED DESCRIPTION:
The aim of this work is therefore the evaluation of Discogel® in the treatment of Discogel®, which appears to be a safe and efficacity of method.

ELIGIBILITY:
Inclusion Criteria:

* Patient with aneurysmal or simple bone cyst who benefit a sclerotherapy by Discogel

Exclusion Criteria:

* Refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with aneurysmal or simple bone cyst who benefit a sclerotherapy by Discogel will be included.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the technique | Year: 2
  Collect from medical records the number of procedures that were completed and performed as theoretically intended.

SECONDARY OUTCOMES:
Safety of the technique by number of adverse event | Year: 2
  collect in the medical record
Number of discogel® injections by sclerose of the lesion | Year: 2
  Efficacity of the technique

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Grange, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No